CLINICAL TRIAL: NCT04605523
Title: Neurofilament Light- Chain as Biomarker for Neurodegeneration in Ataxia Telangiectasia
Brief Title: Neurofilament Light- Chain in Ataxia Telangiectasia
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Stefan Zielen, Head of Pediatric Pulmonology, Johann Wolfgang Goethe University Hospital
Other Study IDs: 168/18
Record Dates: First submitted 2020-10-22; First posted 2020-10-28 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Ataxia Telangiectasia
Keywords: Ataxia telangiectasia; neurodegeneration; biomarker; disease progression; CSF; Neurofilament light chain
MeSH Terms: conditions — Ataxia Telangiectasia; Nerve Degeneration; Disease Progression; Charcot-Marie-Tooth disease, Type 1F

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum of whole blood CSF
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Ataxia Telangiectasia
  Interventions: Procedure: blood withdrawal
- Healthy controls
  Interventions: Procedure: blood withdrawal

INTERVENTIONS:
Procedure: blood withdrawal — Additional blood sample will be taken within blood collection as part of standard care

SUMMARY:
Ataxia telangiectasia (A-T) is a rare autosomal recessive neurodegenerative disorder characterized by progressive cerebellar ataxia, immunodeficiency, chromosomal instability, and cancer susceptibility. Currently there are no curative therapy options. The clinical presentation of the disease has a wide variety is linked to the proven mutation, immunological status and residual ATM kinase activity. Apart from these prognostic markers, hardly any biomarker to predict disease course is available. Aim of the present proposal is to evaluate serum concentrations of neurofilament - light chain in the serum of whole blood as biomarker of neurodegeneration prospectively. In addition to that, the investigators will examine the evolution of neurofilament - light chain longitudinally by blood samples from our biobank as well as the concentration of neurofilament - light chain in cerebrospinal fluid (CSF) of affected A-T patients from our biobank.

As in other neurodegenerative disorders and ataxias, the investigators expect that neurofilament- light chain levels are increased in the A-T cohort and correlated to the neurological status of A-T patients evaluated by means of AT-score.

DETAILED DESCRIPTION:
A-T is a neurodegenerative disease with mutation in the ATM gene. The clinical presentation is complex and affects many different organ systems. Typical findings are progressive cerebellar ataxia, malnutrition, immunodeficiency, chromosomal instability and cancer susceptibility. In addition, new disease entities such as hepatopathy, diabetes and endocrinological alterations are coming to the force.

The severity of the disease is closely related to presence of residual kinase activity, immunological status and specific mutations. However, the individual course of the disease is hard to predict. There is an urgent need to find and define reliable biomarkers for disease progression in order to estimate the prognosis of individual disease course. According the classification of estimated disease severity, the most suitable therapy and support can be organized.

In many other neurodegenerative disorders neurofilament- light chain has been reported to be a sensitive and reproducable serum biomarker for disease progression, activity and monitoring of therapy efficaciousness. Neurofilament proteins indicate neuroaxonal damage independent of causal pathway, the advantage of neurofilaments as a biomarker of disease progression is that levels rise upon neuroaxonal damage not only in CSF but also in blood. Therefore, they can be used to monitor disease activity without invasive procedures.

The aim of the proposal is to measure and evaluate neurofilament-light chain as serum biomarker of disease progression in A-T patients. Additionally, the investigators will measure neurofilament-light chain in CSF from their human biobank and characterize the individual evolution in the serum of whole blood taken from the biobank.

In the prospective part of the study, the investigators will correlate the levels of neurofilament to A-T scores for neurological assessment.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Patients: aged ≥2 and 45 years
* known A-T

Exclusion Criteria:

* cranial trauma in the last 6 months
* ongoing malignant disease
* Chronic diseases or infections (e.g. HIV, Tbc)
* Pregnancy
* Alcohol, substance or drug abuse
* inability to capture extend and consequences of the study

Ages: 2 Years to 45 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients with clinically / and or genetically confirmed diagnosis of ataxia telangiectasia
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Neurofilament - light chain | 01 Feb 2020 - 31 Dec 2020
  Increase of neurofilament between age groups: A: 3-6 years; B: 6- <12 years ; C:12-18 years , D: >18 years. Comparison of absolute levels neurofilament (pg/ml) between groups

SECONDARY OUTCOMES:
Absolute increase per year of neurofilament (pg/ml) | 01 Feb 2020 - 31 Dec 2020
  Absolute increase per year of neurofilament (pg/ml)
Correlation of neurofilament with age | 01 Feb 2020 - 31 Dec 2020
  Correlation of neurofilament with age
Correlation of neurofilament with A-T score | 01 Feb 2020 - 31 Dec 2020
  Correlation of neurofilament with A-T score

OTHER OUTCOMES:
Variability of levels of neurofilament within 12 months | 01 Feb 2020 - 31 Dec 2020
  Variability of levels of neurofilament within 12 months
Levels of neurofilament in cerebrospinal fluid (CSF) | 01 Feb 2020 - 31 Dec 2020
  Levels of neurofilament in cerebrospinal fluid (CSF)
Correlation of neurofilament between serum and CSF | 01 Feb 2020 - 31 Dec 2020
  Correlation of neurofilament between serum and CSF

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Zielen, Prof. Dr., Principal Investigator — University Children´s Hospital, Pediatric Pulmonology
Locations (1):
- University Children´s Hospital, Ped. Pulmonology, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No